CLINICAL TRIAL: NCT06605625
Title: Vaccine Responses in Cancer
Acronym: VRiC
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 852151; UPCC27922 (Other: University of Pennsylvania Cancer Center)
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Viral Vaccines
Keywords: influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Cancer: Patients with cancer who are clinically indicated to receive influenza, recombinant shingles and/or SARS-CoV2 vaccine
  Interventions: Biological: Influenza vaccination; Biological: SARS-CoV-2 vaccine; Biological: Zoster Vaccine Recombinant

INTERVENTIONS:
Biological: Influenza vaccination — one annual dose of inactivated influenza vaccine
Biological: SARS-CoV-2 vaccine — dose of SARS CoV2 vaccine
Biological: Zoster Vaccine Recombinant — first and/or second vaccination for shingles (Herpes zoster)

SUMMARY:
The investigators are conducting a prospective unblinded study of individuals diagnosed with cancer who will receive one or more of the following: influenza, SARS-CoV2 and shingles.

DETAILED DESCRIPTION:
Vaccinations are indicated for all adults, but the immunogenicity of vaccination has not been assessed in all situations. In particular, immune responses following vaccination have not been studied in the setting of cancer and in the context of various anti-tumor treatments. In this study, the investigators will look at the immune response of subjects receiving vaccination.

ELIGIBILITY:
Inclusion Criteria:

* adults over age 18 who are able to provide consent, who have a diagnosis of cancer, and are willing to receive the influenza, recombinant shingles, and/or SARS-CoV-2 vaccines.

Exclusion Criteria:

* allergic to influenza, shingles, and/or SARS-CoV-2 vaccination; have HIV infection; have a history of solid organ or bone marrow transplant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer who are clinically indicated to receive influenza, recombinant shingles (Shingrix) and/or SARS-CoV-2 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody response | 45-90 days
  The neutralizing antibody titer will be assessed by measurement of the hemagglutinin-inhibition titer before and after influenza vaccination in order to determine the seroconversion rate. The late blood draw may occur between days 45-90 following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: E. John Wherry, PhD, Principal Investigator — Univeristy of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No